CLINICAL TRIAL: NCT04098627
Title: The Effects of Laughter Therapy on Hemodialysis on Depression: A Pragmatic Randomized Controlled Trial
Brief Title: The Effects of Laughter Therapy on Hemodialysis on Depression
Acronym: LOL-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SIH109_LOLRCT
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: End Stage Kidney Disease
Keywords: laughter; depression; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Laughter; Depression | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistical Analysis Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Once weekly 30-minute long group laughter therapy session for 8 weeks while patients are on dialysis
  Interventions: Behavioral: Laughter Therapy
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Laughter Therapy — Once weekly 30-minute long group laughter therapy session for 8 weeks
  Arms: Intervention

SUMMARY:
End stage kidney disease is associated with increased depression. Laughter is associated with improvement in depression in chronic disease. The study objective was to measure the effect of intradialytic group laughter therapy on anxiety and depression. Pragmatic randomized controlled trial conducted in 10 hemodialysis centers in Northern California. The intervention group received a once weekly 30-minute long group laughter therapy session for 8 weeks. Primary outcome was depression score as measured using the Patient Health Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of end stage kidney disease (ESKD) and currently undergoing hemodialysis at a Satellite Healthcare Hemodialysis Center
* Ability to understand English

Exclusion Criteria:

* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Depression | 8 weeks
  Change in General Anxiety Disorder Scale 2 (GAD -2) in intervention group compared to change in the usual care group. The construct is the screening measure of depression which is calculated by the sum of 2 items on a scale of 0 to 3. A score of 3 or greater for depression is considered positive for screening purposes. The higher the sore the greater the chance of depression risk and thus the worse outcome.

SECONDARY OUTCOMES:
Anxiety | 8 weeks
  Change in the anxiety subscale of the Patient Health Questionnaire 4 (PHQ4) in intervention group compared to change in the usual care group.The construct is the screening measure of anxiety which is calculated by the sum of 2 items on a scale of 0 to 3. A score of 3 or greater for anxiety is considered positive for screening purposes. The higher the sore the greater the chance of anxiety risk and thus the worse outcome.
Subjective Wellbeing | 8 weeks
  Change in Subjective Wellbeing using the 7 item Personal Wellbeing Index (PWI) in the intervention group compared to change in the usual care group. Subjective wellbeing measures the construct of long term happiness. The Personal Wellbeing Index (PWI) is a 7 item validated scale that rates satisfaction with life in seven domains: standard of living, health, achievements in life, relationships, safety, community and future security, on an 11-point scale. The higher the rating the better the outcome. Measures are individually scored and cumulatively scored.
Patient reported outcome measures (PROMs) | 8 weeks
  Change in PROMS using the 6 item London Evaluation of Illness (LEVIL) in the intervention group compared to change in the usual care group. LEVIL is a 6 item visual analogue scale (VAS) developed and used in hemodialysis patients that measures general wellbeing (GWB), pain, sleep, breathing, energy, and appetite. The anchors for GWB, sleep and appetite were "very poor"-"excellent," for pain and breathing "extreme"-"no problem" and for energy "extremely fatigued"-"full of energy." For each domain the VAS allowed free selection of status along a line from worst (0) to best (100). Measures are individually scored and cumulatively scored.
Psychological Distress - Patient Health Questionnaire 4 (PHQ4) | 8 weeks
  Change in Psychological Distress, as measured by the Patient Health Questionnaire 4 (PHQ4), in intervention group compared to change in the usual care group. The construct is the screening measure of psychological distress which is calculated by the sum of 4 items on a scale of 0 to 3. A score of 0 to 2 is no distress, 3-5 is mild distress, 6-8 is moderate distress and 9-12 is severe distress. The higher the sore the greater the psychological distress and thus the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paul N Bennett, PhD, Principal Investigator — Satellite Healthcare
Locations (1):
- Satellite Healthcare, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No
We plan to keep all data confidential unless requested by statutory body.